CLINICAL TRIAL: NCT04697719
Title: DISCOVER: A Single-site Double-blind Placebo-controlled Randomized Mechanistic Crossover Trial to Assess the Influence of boDy weIght on aSpirin-triggered speCialized prO-resolVing mEdiatoRs
Brief Title: Body Weight, Aspirin Dose and Pro-resolving Mediators
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 20-01884
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Body Weight
Keywords: Aspirin
MeSH Terms: conditions — Body Weight | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: This is a two-phase crossover design with run-in and wash out periods prior to each phase.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aspirin 81mg, Then Aspirin 325mg (Experimental): After a 3 week placebo run-in period, participants first receive Aspirin 81mg capsule daily for 3 weeks. After a placebo washout period of 3 weeks, they then receive Aspirin 325mg capsule daily for another 3 weeks.
  Interventions: Drug: Aspirin 81mg; Drug: Aspirin 325mg
- Aspirin 325mg, Then Aspirin 81mg (Experimental): After a 3 week placebo run-in period, participants first receive Aspirin 325mg capsule daily for 3 weeks. After a placebo washout period of 3 weeks, they then receive Aspirin 81mg capsule daily for another 3 weeks.
  Interventions: Drug: Aspirin 81mg; Drug: Aspirin 325mg

INTERVENTIONS:
Drug: Aspirin 81mg — 81mg oral capsule
Drug: Aspirin 325mg — 325mg oral capsule

SUMMARY:
This study employs a placebo-controlled randomized cross-over design to investigate the impact of body weight and aspirin dose on levels of specialized pro-resolving lipid mediators in blood and neutrophils.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 70 years

Exclusion Criteria:

1. Anti-platelet medication use in the past 7 days
2. Aspirin intolerance or allergy
3. Known bleeding or clotting disorder
4. Chronic inflammatory or connective tissue disease
5. Immunological deficiency
6. Diabetes mellitus
7. Prior gastric or bariatric surgery
8. Active smoking
9. Platelet count <100,000
10. Use of omega-3 fatty acid supplementation
11. Use of drugs or supplements known to inhibit COX-1/COX-2/lipoxygenases
12. Corticosteroid use
13. Recent initiation or change in dose of statin therapy
14. Pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Change in Serum 15R-LXA4 | Week 3, Week 6
Change in Serum 15R-LXA4 | Week 9, Week 12

SECONDARY OUTCOMES:
Change in lipid mediator profile of specialized pro-resolving mediators (SPMs) | Week 3, Week 6
Change in lipid mediator profile of specialized pro-resolving mediators (SPMs) | Week 9, Week 12
Change in lipid mediator profile of leukotrienes | Week 3, Week 6
Change in lipid mediator profile of leukotrienes | Week 9, Week 12
Change in lipid mediator profile of prostaglandins | Week 3, Week 6
Change in lipid mediator profile of prostaglandins | Week 9, Week 12
Change in platelet-monocyte aggregates | Week 3, Week 6
Change in platelet-monocyte aggregates | Week 9, Week 12
Change in platelet-neutrophil aggregates | Week 3, Week 6
Change in platelet-neutrophil aggregates | Week 9, Week 12
Change in platelet surface expression of CD62P | Week 3, Week 6
Change in platelet surface expression of CD62P | Week 9, Week 12
Change in leukocyte expression of ALX/FPR2 | Week 3, Week 6
Change in leukocyte expression of ALX/FPR2 | Week 9, Week 12
Change in leukocyte expression of GPR32 | Week 3, Week 6
Change in leukocyte expression of GPR32 | Week 9, Week 12
Change in leukocyte expression of ERV1/ChemR23 | Week 3, Week 6
Change in leukocyte expression of ERV1/ChemR23 | Week 9, Week 12
Change in leukocyte expression of BLT1 | Week 3, Week 6
Change in leukocyte expression of BLT1 | Week 9, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Sean Heffron, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to sean.heffron@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT04697719/ICF_000.pdf